CLINICAL TRIAL: NCT02088762
Title: Impact of the Excision of Melanoma > 2mm in Thickness With 1cm Surgical Margins on Survival of the Patients in Comparison to 2 cm Surgical Margins
Brief Title: Impact of Excision Margins on Survival and Recurrence Rate in Patients With Thick Melanoma (>2mm)
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 24-08-10
Record Dates: First submitted 2014-03-11; First posted 2014-03-17 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Melanoma
Keywords: margin of safety
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 cm safety margin: 1 cm safety margin
  Interventions: Procedure: surgical excision
- 2 cm safety margin: 2 cm safety margin
  Interventions: Procedure: surgical excision

INTERVENTIONS:
Procedure: surgical excision — comparison of safety margin 1 versus 2 cm

SUMMARY:
Objective: To investigated the impact of the excision of melanoma 2mm≤ in thickness with 1cm surgical margins on survival of the patients compared with 2 cm surgical margins.

Background: Early recognition and appropriate excision play a crucial role in management of malignant melanoma, while the size of surrounding normal skin that should be excised is area of controversies.

Methods: The investigators will conduct a retrospective population-based survey in patients with primary melanoma 2 mm≤ in thickness undergoing tumor excision with 1 cm and 2 cm margins in the investigators center. For both groups, the patients' charts reviewed for data including patient gender, age, tumor location, tumor type, Clark's level, Breslow thickness, tumor type, presence of ulceration, findings of sentinel nodes, local recurrences, locoregional metastases, disease free survival and overall survival were calculated for both groups.

DETAILED DESCRIPTION:
Background

Early recognition and appropriate excision play a crucial role in management of malignant melanoma, while the size of surrounding normal skin that should be excised is area of controversies.

Objective

To investigated the impact of the excision of melanoma 2mm≤ in thickness with 1cm surgical margins on survival of the patients compared with 2 cm surgical margins.

Methods

The investigators will conduct a retrospective population-based survey in patients with primary melanoma 2 mm≤ in thickness undergoing tumor excision with 1 cm and 2 cm margins in the investigators center. For both groups, the patients' charts reviewed for data including patient gender, age, tumor location, tumor type, Clark's level, Breslow thickness, tumor type, presence of ulceration, findings of sentinel nodes, local recurrences, locoregional metastases, disease free survival and overall survival were calculated for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed melanoma
* Safety margin 1 cm or 2 cm
* Tumor thickness according to Breslow >2mm

Exclusion Criteria

* Safety margin less 1 cm
* Unclear safety margins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with melanom of a tumourthickness above 2 mm admitted to the University Hospital of Bern, Inselspital
Sampling Method: Probability Sample
Enrollment: 325 (Actual)
Dates: Start 1997-01; Primary Completion 2012-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | Up to 216 months

SECONDARY OUTCOMES:
Recurrence free survival | Up to 216 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Hunger, MD-PhD, Principal Investigator — Department of Dermatology, University of Bern
Locations (1):
- Department of Dermatology, Bern, Switzerland